CLINICAL TRIAL: NCT05434325
Title: Therapeutic Evaluation of STeroids in IgA Nephropathy Global - Post-Trial ObservatioNal Cohort Study
Brief Title: TESTING -ON Post-Trial ObservatioNal Cohort Study
Acronym: TESTING-ON
Status: Recruiting | Type: Observational
Sponsor: The George Institute (Other)
Collaborators: Peking University Institute of Nephrology (Unknown)
Responsible Party: Sponsor
Other Study IDs: TESTING-ON
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: IgA Nephropathy; ESRD; Glomerulonephritis; Kidney Diseases
Keywords: kidney
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Failure, Chronic; Glomerulonephritis; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TESTING Particpants: All participants who were successfully randomised to the TESTING study who are still alive and have not reached kidney failure requiring dialysis.

SUMMARY:
The primary aim of this study is to extend follow up of TESTING study participants and to assess the long-term effects of a 6-9-month course of oral methylprednisolone on End Stage Kidney Disease (ESKD), according to dose (full-dose vs reduced-dose), ethnicity (Chinese vs other) and kidney function (eGFR above and below 60 mL/min/1.73m2).

DETAILED DESCRIPTION:
In the original TESTING study, the median follow-up for full vs reduced dose cohort was 6.1 vs 2.5 years. We learned from the TESTING trial that the composite endpoints (ESKD, 40% reduction in eGFR or death due to kidney disease) tend to start occurring 2-3 years after randomization. At the time of overall study completion, most of the reported endpoints had occurred in participants from the initial, full-dose TESTING cohort. Although we found the effect of corticosteroid is consistent in both doses, longer follow up is required to confirm the beneficial effects on clinically important renal outcomes of the apparently safer reduced reduced-dose cohort, and to confidently compare the effects across doses. As the trial is assessing the effects of a time-limited 6-9-month period of steroids, a post-trial observation cohort study is a critical, cost and resource-efficient method of answering a number of key questions:

1. Is the apparent benefit of glucocorticoid sustained over long term follow-up?
2. Does a lower dose of steroids safely produce similar benefits on long-term kidney outcomes?

The primary aim of TESTING-ON is to extend follow up of TESTING study participants and to assess the long-term effects of a 6-9-month course of oral methylprednisolone on end stage kidney disease (ESKD), according to dose (full-dose vs reduced-dose), ethnicity (Chinese vs other) and kidney function (eGFR above and below 60 mL/min/1.73m2).

The working hypothesis of TESTING-ON is that a 6-9-month course of oral methylprednisolone will lead to persistent benefits over a long period of time.

TESTING-ON is a post-trial observational study of those participants randomized into the TESTING trial who are still alive, haven't reached ESKD and didn't withdraw consent during the trial. Follow-up will continue for up to five years, with further ongoing follow-up should funding allow.

ELIGIBILITY:
Inclusion Criteria:

1) Only participants who were randomised into the TESTING trial

Exclusion Criteria

1. Participants who have reached kidney failure requiring maintenance dialysis or kidney transplantation during the TESTING trial
2. Participants who died during the TESTING trial
3. Participants who had withdrawn their consent during the TESTING trial
4. Participants who are unable to provide consent for some other reason

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study will consist of all TESTING participants who do not meet any of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 366 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Primary AIM | Through study completion, an average of 1 year
  The development of end stage kidney disease (ESKD) defined as a need for maintenance dialysis or kidney transplantation, and death due to kidney disease

SECONDARY OUTCOMES:
Secondary Aims | Through study completion, an average of 1 year
  The composite of ESKD, 30% decrease in eGFR and all cause death
Secondary Aims | Through Study completion, an average of 1 year
  The composite of ESKD, 40% decrease in eGFR and all cause death
Secondary Aims | Through Study Completion, an average of 1 year
  The composite of ESKD, 50% decrease in eGFR and all cause death
Secondary Aims | Through Study Completion, an average of 1 year
  Each of ESKD, death due to kidney disease and all cause death
Secondary Aims | Through Study Complication an average of 1 Year
  Annual eGFR decline rate
Secondary Aim | Through Study Completion an average of 1 year
  Time averaged proteinuria post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Prof, Study Chair — Peking University Institute of Nephrology; Vlado Perkovic, Prof, Study Chair — University of New South Wales; Muh Geot Wong, Dr, Principal Investigator — University of New Souht Wales; Jicheng Lv, Principal Investigator — Peking University of Nephrology
Locations (58):
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Canada (8):
  - University of Calgary/Alberta Health Services, Calgary, Alberta
  - University of Alberta Hospitals, Edmonton, Alberta
  - St Pauls Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamiliton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital,, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- China (35):
  - Chinese PLA General Hospital (301 Hospital), Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital, Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology,, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Jilin Province FAW General Hospital [Jilin University Fourth Hospital], Changchun, Jilin
  - he First Affiliated Hospital of Dalian Medical University, Dalian, Dalian, Liaoning
  - Shengjing Hospital Of China Medical University, Shengyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Shangdong First Medical University,Shangdong Provincial Qianfoshin, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - The Second Hospital of Shanxi Medical University, Taiyuan, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Science, Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University of Medicine, Hangzhou, Zhejiang
  - Hangzhou Hospital of Traditional Chinese Medicine,, Hangzhou, Zhejiang
  - Ningbo Urology & Nephrology Hospital, Ningbo, Zhejiang
  - Zhejiang Provincial People's Hospital, Sangzhou, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - XinQiao Hospital, Third Military Medical University, Chongqing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University, School of Medicine, Shanghai
- Princess Margaret Hospital, Kowloon, Hong Kong
- India (5):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Nizams Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Calicut Medical College, Kozhikode, Kerala
  - Post Graduate Institue of Medical Education and Reasearch, Chandigarh, Punjab
  - Madras Medical College, Chen, Tamil Nadu
- Malaysia (6):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Kuala Lumpur, Kuala Lumpur, Kulala Lumpur
  - Hospital Tuanku Jaafar Seremban, Seremban, Negri Seremban
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Umum Sarawak, Kuching, Samarahan
  - University Malaysia Medical Centre, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No